CLINICAL TRIAL: NCT07391748
Title: Efficacy of a Polyhexanide Biguanide-Based Gel in the Prevention of Biofilm Formation in Pressure Ulcers
Acronym: EGELPUPP
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Alma Balaguer Menchero, Principal Investigator Alma Balaguer Menchero, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 20250929
Record Dates: First submitted 2025-09-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pressure Ulcers; Pressure Ulcers Stage III; Pressure Ulcer Prevention; Pressure Ulcer ( Stage 2-3); Biofilm Formation; Biofilm; Biofilm Removal
Keywords: Pressure ulcers; biofilms; primary prevention; antimicrobial agents
MeSH Terms: conditions — Pressure Ulcer | interventions — Biguanides; Single Person; Alginates; Silver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gel polihexanida- biguanida Factor (Active Comparator)
  Interventions: Combination Product: To determine the efficacy of a gel containing polyhexanide and biguanide, alone or in combination with alginate with or without silver, in preventing biofilm in PU, in terms of healing at 4 weeks
- Hydrofiber of hydrocolloid with silver (Ag) (Active Comparator)
  Interventions: Combination Product: To determine the efficacy of a gel containing polyhexanide and biguanide, alone or in combination with alginate with or without silver, in preventing biofilm in PU, in terms of healing at 4 weeks

INTERVENTIONS:
Combination Product: To determine the efficacy of a gel containing polyhexanide and biguanide, alone or in combination with alginate with or without silver, in preventing biofilm in PU, in terms of healing at 4 weeks — The intervention consists of the topical application of a gel containing polyhexanide and biguanide (Prontosan®), either alone or in combination with a silver-containing alginate dressing (Aquacel Ag+®), specifically for category II and III pressure ulcers.
  Its efficacy in preventing bacterial biofilm formation in the wound bed and its impact on healing over a four-week period are being evaluated, following the TIME algorithm for wound bed preparation.
  The study employs a 2×2 factorial design, with four treatment groups (gel alone, silver dressing alone, combination of both, and control), and uses standardised assessment tool RESVECH 2.0 to monitor wound progression.

SUMMARY:
INTRODUCTION: Pressure ulcers (PU) are one of the main challenges for nursing in our country. Wound bed preparation and the TIME algorithm provide essential tools for adequately treating these lesions. However, these wounds tend to become chronic due to the bacterial load in their bed. It is now known that bacteria can form complex and diverse structures, named as biofilm, which are difficult to diagnose and much more resistant to antimicrobial action.

Controlling these biofilms is crucial to create the optimal conditions for wound healing. Currently, it is believed that biofilms are present in 60-100% of chronic wounds. Therefore, more studies are needed to evaluate the efficacy of different antimicrobial agents on these structures.

OBJECTIVE: To determine the efficacy of a gel containing polyhexanide and biguanide, alone or in combination with alginate with or without silver, in preventing biofilm in PU, in terms of healing at 4 weeks.

METHODOLOGY: Multicenter clinical trial with a 2x2 factorial design, conducted with patients from Alcoy with category II and III PUs that meet the inclusion and exclusion criteria. A sample of 140 participants is estimated, distributed into four groups of 35 patients. The interventions that will be carried out will be: application of Prontosan gel® and Aquacel Ag+®; Aquacel Ag+®; control group; Prontosan gel®. Data on wound evolution will be collected using RESVECH 2.0. Descriptive statistical analysis and hypothesis testing will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Bedridden patients, patients with bed-to-chair mobility, or those in a wheelchair.
* Presenting one or more category II-III pressure ulcers.
* Aged over 65 years.
* Patients with laboratory results within normal metabolic values (HbA1c < 7%).
* Patients who, in item 6 "infection/suspected biofilm" of the RESVECH 2.0 index, do not have tissue compatible with biofilm, hypergranulation, or purulent exudate, and never score more than 4 in the other items.
* During follow-up, cases that develop signs and symptoms of local infection according to TILI and/or the RESVECH 2.0 index will be considered therapeutic failures, allowing for clinical rescue, but the patient will remain in the intention-to-treat (ITT) analysis.

Exclusion Criteria:

* Patients who, despite the above, present a deteriorated health status that could influence the outcome, such as terminally ill patients, oncology patients, or those with inflammatory diseases.
* Patients in a state of malnutrition according to the Mini Nutritional Assessment (MNA®) scale who are not receiving nutritional supplements, and/or at risk of malnutrition with nutritional deficits.
* Patients with pressure ulcers in the perineal area and urinary incontinence (except those with a urinary catheter) and/or fecal incontinence.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in RESVECH 2.0 score at four weeks in patients with category II and III pressure ulcers treated with polyhexanide-biguanide gel alone or combined with alginate dressing with or without silver, compared with standard care. | From enrollment to the end of treatment at 4 weeks